CLINICAL TRIAL: NCT02389387
Title: Reducing Disparities in Access to Kidney Transplantation: The RaDIANT Regional Study
Brief Title: Reducing Disparities in Access to Kidney Transplantation (RaDIANT) Regional Study
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Rachel Patzer, Assistant Professor, Emory University
Other Study IDs: IRB00079596; 5U01MD010611-05 (NIH)
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: End-stage Renal Disease
Keywords: Dialysis Facilities; African Americans; Racial Disparity; Kidney Transplantation; Community-based Participatory Research; Coalition
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Two hundred twenty (220) dialysis facilities will follow standard of care practices in their management of ESRD patients. They will not receive interventions, but they will have access to standard educational materials and quality improvement through End Stage Renal Disease Network 6.
- Intensive Intervention: Two hundred twenty (220) dialysis facilities will follow standard of care practices and the intensive intervention in their management of ESRD patients. The intensive intervention will consist of 1) A multi-module, secure, web-enabled software application called Transplant Referral EXchange (T-REX) to enhance coordination between dialysis and transplant staff and track ESRD patients through the seven primary steps to transplant , 2) educational webinars/seminars for staff, 3) facility-specific performance feedback reports, 4) assistance with and review of center-specific action plans to increase transplant referral, 5) scheduled bi-annual phone calls with an SETC member to monitor progress, 6) patient education on transplant via creation of an Education Station in facility lobby, and 7) development of a Peer Mentor program.
  Interventions: Other: Intensive Intervention

INTERVENTIONS:
Other: Intensive Intervention — I.A multi-module, secure, web-enabled software application called Transplant Referral EXchange (T-REX):1) real-time communication between staff across healthcare settings, documenting the use of transplant education materials, 2) sending/receiving electronic referrals for transplant specific to a transplant center's requirements and 3) tracking patients' status in the transplant process (e.g., patient interest in transplant, referral for transplant, evaluation start/completion, waitlist status, and transplant) II. Educational webinars/seminars for staff, III. Facility-specific performance feedback reports, IV. Assistance with and review of center-specific action plans to increase transplant referral, V. Scheduled bi-annual phone calls with an SETC member to monitor progress, VI. Patient education on transplant via creation of an Education Station in facility lobby, VII. Development of a Peer Mentor program.
  Groups: Intensive Intervention

SUMMARY:
The purpose of this study is to facilitate coordination of transplant centers in North Carolina, South Carolina, and Georgia to share kidney transplant referral data in patients with End-Stage Renal Disease (ESRD) who are candidates for kidney transplantation.

DETAILED DESCRIPTION:
Disparities exist in access to kidney transplantation where poor and minority patients are less likely to access each step of the kidney transplant process. Current national surveillance data does not capture information on transplant referral, and it is unclear to what extent dialysis facility-level factors may influence disparities in access to transplantation. Due to significant variability in the standardized transplant ratios observed at each facility, the investigators hypothesize that there may be facility-related reasons that impact disparities in access to the first step of the kidney transplant process -- referral to the transplant center to undergo an evaluation for the suitability for transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Kidney transplant centers in the geographic area of North Carolina (NC), South Carolina (SC) and Georgia (GA)
2. Low rates of referral for kidney transplantation (6-month crude referral risk mean of 0.06 and all facilities with a crude referral risk less than the mean)
3. The presence of a racial disparity (African American vs. Caucasian) in referrals for kidney transplantation (racial disparity calculated based on the crude referral risk difference and the standardized referral risk difference.)

The final pool of 440 facilities will be randomized to either the intervention or control group using a one to one ratio.

Exclusion Criteria:

1. Close out date populated
2. Transplant and hospital-based facility
3. Home dialysis facility
4. Patient census <25
5. >100 miles from nearest transplant center
6. Non-profit facility (except Wake Forest University Dialysis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Research assistants from GA transplant centers will contact ~1500 patients via phone. These are patients that were referred for kidney transplant in 2014 that did and did not start the evaluation process. Verbal consent will be obtained, and then conduct the surveys by phone to ensure that patients with any literacy or visual barriers are included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2015-03; Primary Completion 2020-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Referral Disparity from baseline | Baseline, one year after completion of the intervention
  Assessed by referral disparity ratio: percentage of African American patients over percentage of white patients referred (%AA referred/%white referred) to compare across intervention and control facilities at baseline and one year after completion of the intervention. This is a facility level outcome.

SECONDARY OUTCOMES:
Change in medical evaluation start racial disparity and waitlisting racial disparity | Baseline, 6 months after referral, one year after the start of medical evaluation
  Assessed by the racial disparity ratio (%AA/%white) by facility group (control or experimental) for medical evaluation start within 6 months of referral and placement on the waitlist within 1 year of initiating the medical evaluation. This is a facility level outcome.
Change in number of referrals between Control and Experimental patients from baseline | Baseline, 6 months after referral, one year after referral
  Number of individual-patient referrals within 1 year of dialysis start, medical evaluation start within 6 months among those referred, and waitlisting within 1 year among those who start evaluation, among experimental vs. control patients.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Patzer, PhD, Principal Investigator — Emory University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patzer RE, Buford J, Urbanski M, McPherson L, Paul S, Di M, Harding JL, Katz-Greenberg G, Rossi A, Anand PM, Reeves-Daniel A, Jones H, Mulloy L, Pastan SO; Southeastern Kidney Transplant Coalition. Reducing Disparities in Access to Kidney Transplantation Regional Study: A Randomized Trial in the Southeastern United States. Clin J Am Soc Nephrol. 2024 Dec 13;20(2):256-66. doi: 10.2215/CJN.0000000586. Online ahead of print. PMID 39671258

DOCUMENTS (1):
  • Informed Consent Form (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/87/NCT02389387/ICF_000.pdf